CLINICAL TRIAL: NCT04957641
Title: A Retrospective Observational Chart Review Study Evaluating the Burden of Illness and Treatment Patterns in Hereditary Angioedema Type I and II
Brief Title: A Study of the Burden of Illness and Treatment Patterns in Teenagers and Adults With Hereditary Angioedema
Acronym: BOISTERN
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4009; MACS-2020-080401 (Other: Sponsor)
Record Dates: First submitted 2021-07-05; First posted 2021-07-12 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with HAE: Participants' data will be collected retrospectively from electronic medical records using chart review of de-identified data on participant demographics, HAE medical history and information on diagnostics, treatments and disease course assessments that are routinely performed in accordance with current guidelines and/or local standard of care which are entered into an Electronic data capture (EDC) system over multiple data collection waves up to 6 months.

SUMMARY:
This study is about teenagers and adults with hereditary angioedema (HAE) type I and type II. In this study, the burden of illness means the impact of HAE in terms of long-term health outcomes and the financial cost.

The main aims of this study are as follows:

* to learn how often, how severe and where on the body HAE attacks occur.
* to describe how HAE prophylaxis and on-demand medicines are prescribed and used. (Prophylaxis medicines prevent a bleed from happening and on-demand medicines treat a bleed when it occurs.)

This study is about collecting data only; participants will not receive treatment as part of this study. Existing data available in the participant's medical records will be collected. Participants will be asked to complete an electronic questionnaire either on a website or by using an app on their mobile phone; data from this questionnaire will also be collected.

Participants do not need to visit their doctor in addition to their normal visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged >= 12 years at the time of the last documented HAE attack in the eligibility period.
* Physician-confirmed diagnosis (or confirmation in medical records) of HAE type I or type II.
* Participant had at least one documented HAE attack during the eligibility period.
* Participant is not adequately or sub-optimally controlled according to treating physician.
* Participant (or parent/legal guardian) is willing and able to comply with the study requirements and provides informed consent or assent.

Exclusion Criteria:

* Participant enrolled in a therapeutic investigational drug or device trial during the observation period.
* Participant initiated long-term prophylaxis with Takhzyro® at any time since diagnosis.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged greater than or equal to (>=) 12 years with HAE type I or type II suffering from recurrent attacks will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With HAE Attacks Occurrence During Study Period | Throughout the study period (up to 6 months)
  HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of participants with HAE attacks occurrence (start and end date of each HAE attack) during study period will be reported.
Number of Participants Categorized Based on Characteristics of HAE Attacks During Study Period | Throughout the study period (up to 6 months)
  HAE attack characteristics will be based on prodromal symptoms, severity and location, whether attack was life-threatening will be reported.
Time Interval Between HAE Attacks During Study Period | Throughout the study period (up to 6 months)
  Time interval between HAE attacks during the study period will be reported.
Duration of Each HAE Attacks During Study Period | Throughout the study period (up to 6 months)
  Duration of each HAE attacks during study period will be reported.
Number of Participants Based on Type of HAE Prophylactic Treatments | Throughout the study period (up to 6 months)
  Number of participants based on type of HAE prophylactic treatment will be reported.
Number of Participants Based on Long-term or Short-term HAE Prophylactic Treatment | Throughout the study period (up to 6 months)
  Number of participants based on long-term or short-term HAE prophylactic treatment will be reported.
Number of Participants Categorized Based on Reasons for HAE Prophylactic Treatment Initiation | Throughout the study period (up to 6 months)
  Number of participants categorized based on reasons for HAE prophylactic treatment initiation will be reported.
Duration of HAE Prophylactic Treatment | Throughout the study period (up to 6 months)
  Duration of HAE prophylactic treatment includes treatment start and end dates will be reported.
Number of Participants Categorized Based on Dose and Route of Administration for HAE Prophylactic Treatment | Throughout the study period (up to 6 months)
  Number of participants categorized based on dose and route of administration for HAE prophylactic treatment will be reported.
Number of Participants Categorized Based on Reasons for HAE Prophylactic Treatment Discontinuation | Throughout the study period (up to 6 months)
  Number of participants categorized based on reasons for HAE prophylactic treatment discontinuation will be reported.
Number of Participants Based on Type of HAE On-demand Treatment | Throughout the study period (up to 6 months)
  Number of participants based on type of HAE on-demand treatment will be reported.
Duration of HAE On-demand Treatment | Throughout the study period (up to 6 months)
  Duration of HAE on-demand treatment includes treatment start and end dates will be reported.
Number of Participants Categorized Based on Dose and Route of Administration for HAE On-demand Treatment | Throughout the study period (up to 6 months)
  Number of participants categorized based on dose, route of administration and setting of administration for HAE on-demand treatment will be reported.
Number of Participants Associated Between Prescriptions Patterns and HAE Attacks | Throughout the study period (up to 6 months)
  Number of participants with association between prescriptions patterns and HAE attacks related to frequency or severity. Generalized linear models (GLM) will be used to evaluate the association of outcomes of interest with relevant covariates between prescription pattern, HAE attacks, frequency and severity of HAE attacks will be reported.

SECONDARY OUTCOMES:
Healthcare Resource Utilization (HRU): Number of Visits to Healthcare Professionals (HCP) | Throughout the study period (up to 6 months)
  HRU is measured by the number of visits to HCP will be reported.
HRU: Number of Participants With Emergency Room/Emergency Departments (ER/ED) Visits due to HAE Attacks | Throughout the study period (up to 6 months)
  Number of participants with ER/ED visits due to HAE attacks will be reported.
HRU: Number of Participants With Hospitalizations due to HAE Attacks | Throughout the study period (up to 6 months)
  Number of participants with hospitalizations due to HAE attacks will be reported.
Health-related Quality of Life (HRQoL): Angioedema Quality of Life (AE-QoL) Questionnaire | Throughout the study period (up to 6 months)
  The AE-QoL was developed to measure HRQoL in participants with recurrent angioedema. It is a self-administered patient-reported outcome instrument with a recall period of four weeks. There are 17 items across four domains: functioning (four items), fatigue/mood (five items), fears/shame (six items), and food (two items). Responses use a 5-point Likert scale ranging from 1 (Never) to 5 (Very Often). Global scores range from 0 to 100 and scores by domains range from 0 to 100. An overall score is calculated and a higher score indicates lower quality of life.
HRQoL: EuroQoL Group 5-Dimension 5-Level (EQ-5D-5L) Questionnaire | Throughout the study period (up to 6 months)
  The EQ-5D-5L descriptive system assesses health in five dimensions (Mobility, Self-Care, Usual Activities, Pain / Discomfort, Anxiety / Depression), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). This part of the EQ-5D questionnaire provides a descriptive profile that can be used to generate a health state profile. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the participant rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
HRQoL: EuroQoL-five Dimensions, Youth Version (EQ-5D-Y) | Throughout the study period (up to 6 months)
  The EQ-5D-Y is composed of two sections. The first section contains one question for each of the five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy. Participants select from three response levels (no problems, some problems, a lot of problems) for each dimension. A health state profile score can be calculated from the responses on these five questions. The second section includes the same visual analogue scale as the EQ-5D-5L. The scale is scored from 0-100. The reference to a high score indicates a better outcome of quality of life.
Number of Participants With HAE Attacks Occurrence in Relevant Subgroups | Throughout the study period (up to 6 months)
  HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Relevant subgroups is defined by disease characteristics (e.g., number of attacks) and treatment patterns (type of treatments for HAE). Number of participants with HAE attacks occurrence (start and end date of each HAE attack) in relevant subgroups will be reported.
Number of Participants Categorized Based on Characteristics of HAE Attacks in Relevant Subgroups | Throughout the study period (up to 6 months)
  HAE attack characteristics will be based on prodromal symptoms, severity and location, whether attack was life-threatening in relevant subgroups will be reported. Relevant subgroups is defined by disease characteristics (e.g., number of attacks) and treatment patterns (type of treatments for HAE).
Time Interval Between HAE Attacks in Relevant Subgroups | Throughout the study period (up to 6 months)
  Time interval between HAE attacks in relevant subgroups will be reported. Relevant subgroups is defined by disease characteristics (e.g., number of attacks) and treatment patterns (type of treatments for HAE).
Duration of Each HAE Attacks in Relevant Subgroups | Throughout the study period (up to 6 months)
  Duration of each HAE attacks in relevant subgroups will be reported. Relevant subgroups is defined by disease characteristics (e.g., number of attacks) and treatment patterns (type of treatments for HAE).
HAE Attacks Prescription Pattern in Relevant Subgroups | Throughout the study period (up to 6 months)
  Prescription pattern of HAE attacks medication by drug class in relevant participant subgroups during study period. Relevant subgroups is defined by disease characteristics (e.g., number of attacks) and treatment patterns (type of treatments for HAE).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (36):
- Medizinische Universitat Wien (Medical University of Vienna), Vienna, Austria
- UZ Antwerpen, Edegem, Belgium
- University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia, Bulgaria
- Canada (2):
  - Vancouver Allergy Clinic, Vancouver, British Columbia
  - McMaster University Medical Centre, Hamilton
- Croatia (2):
  - General Hospital Sibenik, Šibenik
  - Klinicki bolnicki centar Zagreb, Zagreb
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice v Motole, Prague
- East Tallinn Central Hospital, Tallinn, Estonia
- Universitätsklinikum Frankfurt, Frankfurt, Germany
- Greece (3):
  - Navy Hospital of Athens, Athens
  - Laiko General Hospital of Athens, Athens
  - University General Hospital of Larissa, Larissa
- Semmelweis Egyetem, Budapest, Hungary
- St James's Hospital, Dublin, Ireland
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Centre of Investigation and Treatment of Allergic Diseases, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Medical Faculty of Ss. Cyril and Methodius Univers, Skopje, North Macedonia
- Wojskowy Instytut Medyczny, Warsaw, Poland
- Portugal (3):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de São João, E.P.E., Porto
- MediQuest Clinical Research Center, Sângeorgiu de Mures, Romania
- University Clinical Center of Serbia - PPDS, Belgrade, Serbia
- Univerzitna nemocnica Martin, Martin, Slovakia
- Bolnisnica Golnik - Klinicni Oddelek za Pljucne Bolezni In Alergijo, Golnik, Slovenia
- Spain (3):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Farkas H, Aygoren-Pursun E, Ebo DG, Bara N, Psarros F, Gavini F, Bent-Ennakhil N, Sayegh L, Andresen I. Real-world treatment patterns and burden-of-disease of sub-optimally controlled hereditary angioedema. World Allergy Organ J. 2025 Sep 1;18(9):101100. doi: 10.1016/j.waojou.2025.101100. eCollection 2025 Sep. PMID 40949786
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60f13b09f883ca001e82d334